CLINICAL TRIAL: NCT02027766
Title: Local and Systemic Changes in Pain Sensitivity After 4 Weeks of Calf Muscle-tendon Stretching: A Randomised Trial
Brief Title: Stretching and Pain Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Senior Researcher, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 129
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Stretching

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Stretching (Experimental): Daily stretching of the calf (dominant side; defined as leg used to kick a ball). 2 stretching exercises are performed daily: 1) stretching of the soleus muscle; 2) stretching of the gastrocnemius muscle.
  Interventions: Other: Calf muscle stretching
- Control (No Intervention)

INTERVENTIONS:
Other: Calf muscle stretching
  Arms: Stretching

SUMMARY:
Stretching is frequently used in clinical practice to manage musculoskeletal discomfort and to prevent sports injuries. It is not known if stretching affects pain sensitivity. The purpose of this study is to investigate if a 4 week daily stretching protocol alters pain sensitivity.

The investigators hypothesize that stretching reduces pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40
* In general good health, in the opinion of the Investigator, based on medical and physical history.
* Speaks, reads and writes Danish language.

Exclusion Criteria:

* Regular use of stretching
* History of surgery to the lower limb(s)
* History of traumatic and overuse injures to the lower limb(s), including but not limited to: Tendinopathies, Bursitis, Muscle injuries, Significant ankle sprains, other ligament injuries
* Hyper mobility syndromes, including but not limited to Ehlers-Danlos syndrome, Generalised hyper mobility syndrome
* History of symptoms of autoimmune disorders (e.g., inflammatory bowel disease, multiple sclerosis, lupus, rheumatoid arthritis).
* Planned surgical procedure during the duration of the study
* History, diagnosis, or signs and symptoms of clinically significant neurological disease, including but not limited to: Stroke or transient ischemic attack, Alzheimer's disease or other types of dementia, Clinically significant head trauma within the past year, Peripheral neuropathy, Epilepsy or seizure, Impaired balance
* Alcohol or drug abuse within the last 5 years
* History, diagnosis, signs or symptoms of any clinically significant psychiatric disorder
* Diabetes
* Subjects with regional pain syndromes suggestive of lumbar compressions with radiculopathy or at risk of developing radiculopathy.
* Any other condition, which in the opinion of the Investigator, would put the subject at increased safety risk or otherwise make the subject unsuitable for this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pressure pain threshold (PPT) at the ipsilateral (same side as being stretched) calf assessed by a cuff pressure algometer | Baseline and after 4 weeks

SECONDARY OUTCOMES:
Change from baseline in PPT at the counter lateral calf | Baseline and 4 weeks
Change from baseline in PPT at the ipsilateral arm | baseline and 4 weeks
Change from baseline in temporal summation of pressure pain at both calfs and ipsilateral arm. | Baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PT, PhD, Principal Investigator — Frederiksberg Hospital
Locations (1):
- The Parker Institute, Bispebjerg and Frederiksberg University Hospitals, Copenhagen, Denmark